CLINICAL TRIAL: NCT05699473
Title: A Double Blind, Randomized, Cross-over, Comparative Bioavailability Study of 3 Different Forms of Folate in Healthy Subjects
Brief Title: Bioavailability Study of Folate in Healthy Subjects
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Analytic issue
Sponsor: Lesaffre International (Industry)
Collaborators: BioFortis (Other); Soladis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PEC21152
Record Dates: First submitted 2023-01-05; First posted 2023-01-26 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-01

CONDITIONS: Healthy
Keywords: folate; bioavailability; comparative study; single dose

STUDY DESIGN:
Intervention Model Description: Prospective, monocentric, double-blind, randomized, cross-over bioavailability study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization list will be drawn up before the beginning of the study by a person not related to the study and stored confidentially. Every effort will be made to maintain the blind during the study.
  The labelling will not show any difference (including batch number and use-by date) between the test and the comparative products.
  During the whole study and in the absence of unblinding, neither the investigators, service providers, nor the participant will be aware of the product they test or can deduce the group they belong to.
  The unblinding will occur after the database locking, at the end of the study. The unblinding will be in charge of the person responsible for the randomization list.
  Whether an emergency unblinding procedure may occur (i.e., SAE), the date and the reason for the unblinding will be indicated in the electronic Case Report Form (e-CRF) and the source document of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 5-MTHF glucosamine (Experimental): 1 single dose (400µg)
  Interventions: Dietary Supplement: 5-MTHF glucosamine salt
- 5-MTHF calcium salt 1 (Experimental): 1 single dose (400µg)
  Interventions: Dietary Supplement: 5-MTHF calcium salt 1
- 5-MTHF calcium salt 2 (Experimental): 1 single dose (400µg)
  Interventions: Dietary Supplement: 5-MTHF calcium salt 2

INTERVENTIONS:
Dietary Supplement: 5-MTHF glucosamine salt — Active form of folate defined as (6S) 5-methyltetrahydrofolate (5-MTHF) glucosamine salt
  Arms: 5-MTHF glucosamine
Dietary Supplement: 5-MTHF calcium salt 1 — Active form of folate defined as (6S) 5-methyltetrahydrofolate (5-MTHF) calcium salt, crystal form 1
  Arms: 5-MTHF calcium salt 1
Dietary Supplement: 5-MTHF calcium salt 2 — Active form of folate defined as (6S) 5-methyltetrahydrofolate (5-MTHF) calcium salt, crystal form 2
  Arms: 5-MTHF calcium salt 2

SUMMARY:
The aim of this prospective interventional study is to compare the bioavailability of the 6S-5-methyltetrahydrofolate (5-MTHF) glucosamine salt versus two other forms of 5- MTHF calcium salts by measuring serum 5-MTHF responses after a single ingestion of equivalent doses of the three folate forms in humans.

The hypothesis of this study is that the test products 5-MTHF glucosamine and calcium salts have equivalent bioavailabilities in serum 5-MTHF as measured by the area under the curve over a period of 24 hours (AUC0-24h) after consumption of a single dose of 5-MTHF (400μg).

Participants will receive a single dose of each of the following products separated by a 7-day wash-out period:

* 5-MTHF glucosamine salt
* 5-MTHF calcium salt 1
* 5-MTHF calcium salt 2

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≥18 and ≤25Kg/m²,
* For women: menopausal without hormone replacement therapy (HRT) or with HRT started from more than 3 months or non-menopausal with a negative blood pregnancy test and using reliable contraception since at least 3 cycles before the beginning of the study and agreeing to keep it during the entire duration of the study,
* Good general and mental health within the opinion of the investigator: no clinically significant and relevant abnormalities of medical history or physical examination,
* Able and willing to participate to the study by complying with the protocol procedures as evidenced by his/her dated and signed informed consent form,
* Affiliated with a social security scheme,
* Agree to be registered on the subjects in biomedical research file.

After V1 biological analysis the subjects will be eligible to the study on the following criteria:

- Adequate folate status (serum folate between 10 and 45nmol/L, erythrocyte (RBC) folate between 405 and 952 nmol/L),

Exclusion Criteria:

* Suffering from a metabolic disorder,
* Suffering from a severe chronic disease found to be inconsistent with the conduct of the study by the investigator,
* Suffering from diseases that could potentially interfere with folate absorption or metabolism,
* With a known or suspected food allergy or intolerance or hypersensitivity to any of the study products' ingredient,
* With a low venous capital of blood samples according to the investigator's opinion,
* Pregnant or was pregnant less than 6 months prior to the study, or lactating women or intending to become pregnant within 3 months ahead,
* Under treatment or regular use of treatment or dietary supplement which could significantly affect folate status or other study parameter(s),
* Use of supplements containing folate (i.e. folic acid, 5-MTHF) the last 3 months,
* With significant change in lifestyle, food habits, physical activity or medications in the 3 months before the V1 visit or not agreeing to keep them unchanged throughout the study,
* With a current or planned in the next 3 months' specific diet (hyper or hypocaloric, vegan, vegetarian…) or stopped less than 3 months before the study,
* With a personal history of anorexia nervosa, bulimia or significant eating disorders according to the investigator,
* Consuming more than 2 standard drinks of alcoholic beverage daily for men and women or not agreeing to keep his alcohol consumption habits unchanged throughout the study.
* Smoking,
* Having a lifestyle deemed incompatible with the study according to the investigator including high level physical activity,
* Taking part in another clinical trial or being in the exclusion period of a previous clinical trial,
* Having received, during the last 12 months, indemnities for clinical trial higher or equal to 4500 Euros,
* Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision,
* Presenting a psychological or linguistic incapability to sign the informed consent,
* Impossible to contact in case of emergency.
* Who made a blood donation in the 3 months before the V0 visit or intending to make it within 3 months ahead.

After V1 biological analysis the subjects will be non-eligible to the study on the following criteria:

* Presence of anemia (hemoglobin<12g/dL in women and 13g/dL in men),
* Vitamin B12 levels (serum cobalamin <148pmol/L),
* Serum total homocysteine levels≥15µmol/L,
* Serum creatinine >0,96mg/dL for women and >1,21mg/dL for men,
* Control record (Glycaemia, total cholesterol, triglycerides, HDL cholesterol, LDL cholesterol, GGT, ASAT, ALAT, Urea and CBC) with clinically significant abnormality according to the investigator.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2023-05-06 (Actual); Study Completion 2023-05-06 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) 0-24 hours of serum 5-MTHF concentrations | 0-24 hours
  Comparison of AUC0-24 hours of serum 5-MTHF concentrations between the 3 study products

SECONDARY OUTCOMES:
Area under the curve (AUC) 0-24 hours of serum total folate concentrations | 0-24 hours
  Comparison of AUC0-24 hours of serum total folate concentrations between the 3 study products
Area under the curve (AUC) 0-8 hours of serum 5-MTHF and total folate concentrations | 0-8 hours
  Comparison of AUC0-8 hours of serum 5-MTHF and total folate concentrations between the 3 study products
Area under the curve (AUC) 0-infinity of serum 5-MTHF and total folate concentrations | 0-24 hours
  Comparison of AUC0-infinity of serum 5-MTHF and total folate concentrations between the 3 study products
Peak plasma concentrations (Cmax) of serum 5-MTHF and total folate | 0-24 hours
  Comparison of peak plasma concentrations (Cmax) of serum 5-MTHF and total folate between the 3 study products
Half-life time of serum 5-MTHF and total folate | 0-24 hours
  Comparison of half-life time of serum 5-MTHF and total folate between the 3 study products
Mean Residence Time (MRT) of serum 5-MTHF and total folate | 0-24 hours
  Comparison of Mean Residence Time (MRT) of serum 5-MTHF and total folate between the 3 study products
Area under the curve (AUC) 0-24 hours of serum 5-MTHF and total folate concentrations adjusted on sex | 0-24 hours
  Comparison of AUC0-24 hours of serum 5-MTHF and total folate concentrations between the 3 study products after adjustment by sex

OTHER OUTCOMES:
Frequency of adverse events (AE) | 4 weeks (inclusion to last visit)
  Frequency of adverse events (AE) occurring during the all duration of the study (AE, serious AE (SAE) and their characteristics (severity, relationship to the research procedure or study product, action taken on the study product, evolution of AE and body system)).
Frenquency of Treatment-Emergent Adverse events (TEAE) | 4 weeks (inclusion to last visit)
  Frequency of Treatment-Emergent Adverse events (TEAE) and their characteristics (severity, relationship to the research procedure or study product, action taken on the study product, evolution of AE and body system).
Frenquency of Serious treatment-emergent adverse events (STEAE) | 4 weeks (inclusion to last visit)
  Frequency of Serious treatment-emergent adverse events (STEAE) and their characteristics (severity, relationship to the research procedure or study product, action taken on the study product, evolution of AE and body system).

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle METREAU, MD, Principal Investigator — BioFortis
Locations (1):
- Biofortis, Saint-Herblain, France

IPD SHARING:
Plan to Share IPD: No